CLINICAL TRIAL: NCT02266069
Title: Implementation of the Care Pathway for Primary Palliative Care in Five Research Clusters in Belgium
Brief Title: PROject - Supportive and Palliative Care and INnOvation - Antwerp (Pro-Spinoza)
Acronym: pro-Spinoza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bert Leysen (Other)
Collaborators: Intermutualistic Agency (Other); National Institute for Health and Disability Insurance, Belgium (Unknown)
Responsible Party: Sponsor-Investigator, Bert Leysen, MD, PhD candidate, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UA C130298
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Palliative Care; Primary Health Care
Keywords: implementation; anticipatory care planning; symptom assessment; interdisciplinary collaboration
MeSH Terms: interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Research cluster 1: Antwerp (Other): The first Dutch-speaking research cluster in a stepped wedge cluster design. Family doctors are implementing the Care Pathway for Primary Palliative Care and will recruit eligible patients from October 2014.
  Interventions: Other: Care Pathway for Primary Palliative Care
- Research cluster 2: Mons (Other): The first French-speaking research cluster in a stepped wedge cluster design. Family doctors are implementing the Care Pathway for Primary Palliative Care and will recruit eligible patients from November 2014.
  Interventions: Other: Care Pathway for Primary Palliative Care
- Research cluster 3: Brussels (Other): The only bilingual Dutch/French-speaking research cluster in a stepped wedge cluster design. Family doctors are implementing the Care Pathway for Primary Palliative Care and will recruit eligible patients from December 2014.
  Interventions: Other: Care Pathway for Primary Palliative Care
- Research cluster 4: Limburg (Other): The second Dutch-speaking research cluster in a stepped wedge cluster design. Family doctors will implement the Care Pathway for Primary Palliative Care and will recruit eligible patients from April 2015.
  Interventions: Other: Care Pathway for Primary Palliative Care
- Research cluster 5: ? (Other): A second French-speaking research cluster in a stepped wedge cluster design. Family doctors will implement the Care Pathway for Primary Palliative Care and will recruit eligible patients from October 2015.
  Interventions: Other: Care Pathway for Primary Palliative Care

INTERVENTIONS:
Other: Care Pathway for Primary Palliative Care — Early identification of palliative care patients, anticipatory care planning, systematic symptom assessment, interdisciplinary collaboration, rigorous follow-up of the functional status of the patient and giving attention to the informal care givers.
  Other Names: CPPPC

SUMMARY:
It is important to provide high quality palliative care to all patients with a non-curable and life-limiting condition. The Care Pathway for Primary Palliative Care (CPPPC) provides tools for health care professionals to help them delivering palliative care timely and accurately.This study investigates whether the implementation of the CPPPC really helps to improve patients' lifes.

ELIGIBILITY:
Inclusion Criteria:

* identified as a palliative care patient using the Surprise Question "Would you, as a family doctor, be surprised if this patient would die in the next 12 months?". If the answer is 'no', the patient is eligible for the study.

Exclusion Criteria:

* not having signed the informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
percentage of deaths occurred in the hospital (of patients per family doctor/per research cluster) | 6 months
  The hypothesis is that the CPPPC reduces the percentage of deaths occurred in the hospital

SECONDARY OUTCOMES:
cost of health care consumption in the last year of life (of patients per family doctor/per research cluster) | 6 months
  The hypothesis is that the CPPPC reduces the cost of health care consumption in the last year of life
consumption of antibiotics in the last year of life (of patients per family doctor/per research cluster) | 6 months
  The hypothesis is that the CPPPC reduces the consumption of antibiotics in the last year of life
consumption of pain killers in the last year of life (of patients per family doctor/per research cluster) | 6 months
  The hypothesis is that the CPPPC augments the consumption of pain killers in the last year of life
consumption of (invasive) diagnostic and therapeutic procedures in the last year of life (of patients per family doctor/per research cluster) | 6 months
  The hypothesis is that the CPPPC reduces the consumption of (invasive) diagnostic and therapeutic procedures in the last year of life

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van den Eynden, MD, PhD, Principal Investigator — Universiteit Antwerpen; Johan Wens, MD, PhD, Principal Investigator — Universiteit Antwerpen
Locations (4):
- Belgium (4):
  - Reliance, Mons, Hainaut
  - Netwerk Palliatieve Zorg Limburg, Hasselt, Limburg
  - Palliatieve Hulpverlening Antwerpen, Antwerp
  - Palliabru, Brussels-Capital Region

REFERENCES:
- [Derived] Leysen B, Van den Eynden B, Janssens A, Wens J. Recruiting general practitioners for palliative care research in primary care: real-life barriers explained. BMC Fam Pract. 2019 Mar 5;20(1):40. doi: 10.1186/s12875-019-0930-y. PMID 30836994
- [Derived] Leysen B, Van den Eynden B, Gielen B, Bastiaens H, Wens J. Implementation of a Care Pathway for Primary Palliative Care in 5 research clusters in Belgium: quasi-experimental study protocol and innovations in data collection (pro-SPINOZA). BMC Palliat Care. 2015 Sep 28;14:46. doi: 10.1186/s12904-015-0043-x. PMID 26416574
- See also: Related Info — http://www.pro-spinoza.be